CLINICAL TRIAL: NCT04025814
Title: A Digital Health Solution for Improving Parent Adherence to Behavioral Treatment for ADHD
Brief Title: dHealth Solution for Improving Parent Adherence to Behavioral Treatment for ADHD
Acronym: dHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-28558
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- dHealth tool and BPT Group (Experimental): Parents and School Mental Health Providers (SMHPs) will participate in a 2-month trial during which they will use a digital Health (dHealth) tool in daily life contexts while receiving BPT, aimed to improve parent adherence sustained use of evidence-based parenting strategies. They will also participate in focus groups and discussions to facilitate the build, design, and use of the dHealth.
  Interventions: Device: CaregiverAssist; Behavioral: Behavioral Parent Training (CLS Parent Group)
- BPT Group (Experimental): Parents and School Mental Health Providers (SMHPs) will participate in a 2-month trial during which they will be receiving BPT without the use of a digital Health (dHealth) tool.
  Interventions: Behavioral: Behavioral Parent Training (CLS Parent Group)

INTERVENTIONS:
Device: CaregiverAssist — CaregiverAssist is a proposed dHealth tool to promote parent adherence and sustained strategy use of evidence-based parenting strategies.
  Arms: dHealth tool and BPT Group
Behavioral: Behavioral Parent Training (CLS Parent Group) — Collaborative Life Skills (CLS) program is implemented at school sites by school mental health providers who are trained by University of California San Francisco (UCSF) project staff

SUMMARY:
This study aims to develop, refine and preliminarily test a novel and scalable digital health solution designed to address parent adherence barriers in daily life contexts and increase parent's sustained use of evidence-based parenting strategies.

DETAILED DESCRIPTION:
The study includes the following 3 phases:

1. Discovery phase: During the Discovery phase, we will conduct 1-hour focus groups at school sites with parents (N=8) and school mental health providers (N=4), who are considered major stakeholders and potential users of the dHealth tool. The purpose of these groups is to obtain feedback and guidance on features and procedures in order to maximize the usability and feasibility of the dHealth tool. This design includes participants who have completed a parenting skills treatment (CLS) and thus would be better informed to comment on needs for the augmented treatment. Stakeholders will be queried about their preferences regarding the application layout, tools, content, and features (e.g., reminders, badges). Recorded focus group sessions will be transcribed and coded for themes related to usability and feasibility.
2. Design and Build phases: Feedback from the discovery phase will be incorporated into the design and build phases, during which time prototypes will be put through proof of concept testing with parents and school clinicians who had participated in the discovery phase. Qualitative data will be collected at 2 time points during the design and build phases. Quantitative data will be gathered using the System Usability Scale (SUS) for each component prototype (e.g., description of skill, video examples, interactive activities). A fully functioning application will be completed at the end of the build phase and ready for the test phase.
3. Test Phase: The test phase is a 2-month pilot open trial of the dHealth tool with parents. We will provide the dHealth tool to parents who participated in the prior phases (N=5) as well as a new sample of parents (N=12) who will test the tool with their children in conjunction with the parent's participation in BPT at their school (to test tool utility during the course of treatment). Parents will be advised to use the tool daily to record parenting strategy use and to access information/training as needed. Qualitative semi-structured interviews during and after the trial will assess reactions to the platform (usability, feasibility, acceptability) to inform refinements and identify barriers and facilitators relating to use. Primary outcomes focus on usage metrics with the tool (e.g., frequency of use, module and activity completion, time, repeat activity), reported daily parenting skills use on the tool, and measures of feasibility and acceptability. Application usage analytics will be collected by the mobile application, providing objective descriptives including how often and for how long individuals access the application and each component, as well as how users navigate through the application. This data will be analyzed for patterns associated with tool satisfaction ratings, feasibility, and acceptability ratings and reported skill utilization. Secondary outcomes of parent knowledge, motivation and confidence in using EBT skills; parenting practices, ADHD symptoms and functional outcomes will be assessed before and after tool usage.
4. Randomized Controlled Trial (RCT) Phase: The RCT phase is a 20-month pilot randomized controlled trial of the refined dHealth tool with parents. We will randomly assign groups to receive either the parenting skills training plus the tool (N=5 groups, 30 parents) or parenting skills training without the tool (N=5 groups, 30 parents). Exploratory analyses will examine the potential mediating mechanism of skill utilization (immediate and sustained) for optimizing the association between the dHealth intervention and improved child and parenting outcomes and the potential moderating effect of parent ADHD/EF functioning and internalizing mental health dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-11 (grades 1-5)
* Identification by school mental health professionals as experiencing challenges with inattention and/or hyperactivity/impulsivity
* Attending a participating SFUSD elementary school full time in a mainstream classroom
* Living with a caretaker who is available to participate in treatment
* Absence of significant visual/hearing impairment, severe language delay, psychosis, pervasive developmental disorder, or global intellectual impairment per school records
* Significant ADHD symptoms as evidenced by having (i) six or more symptoms of inattention and/or hyperactivity/impulsivity rated as occurring "often" or "very often" by parents, (ii) at least one area of functioning rated as -≥ 3 on the Impairment Rating Scale by parent

Exclusion Criteria:

* No presence of conditions that are incompatible with this study's treatment including: severe visual or hearing impairment, severe language delay or intellectual impairment, psychosis, pervasive developmental disorder,
* Child is in an all-day special education classroom (children in these classrooms are frequently receiving intensive behavior modification programs such that the intervention would be expected to require modification for use in these settings)
* Children planning to change (start or stop) psychotropic medication Note: Children taking medication will be required to meet all entry criteria, including impairment criteria, thus indicating a need for the intervention. Children taking medication for attention or behavior are eligible as long as their medication regimens are stable.

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | Change from baseline on technology usability at 6 months
  10-item sale for assessing technology product usability
Feasibility Rating Scale | Change from baseline on technology use at 6 months
  1-5 Likert scale rating of amount of time and level of effort needed to use the tool regularly
Parent Acceptability and Satisfaction Questionnaire | Change from baseline on technology use at 6 months
  1-5 Likert scale rating level of engagement, usefulness, and acceptability
Parent adherence/implementation | Change from baseline on application use at 2 months
  5-point Likert scale rating daily use of skills and behavior plans (tracked on application)

SECONDARY OUTCOMES:
Parent Confidence and Motivation to Use Evidence Based Parenting Skills | Change from baseline on confidence and motivation at 2 months
  5-point Likert scale of parent rated confidence and motivation
Parent Knowledge of Evidence Based Parenting Skills | Change from baseline on knowledge of EBT at 2 months
  Assessed via content question, vignettes, and behavior plans to rate parent knowledge of EBT skills
Alabama Parenting Questionnaire | Change from baseline on parenting skills at 2 months
  Assessment of parenting skills
Parenting Stress Index | Change from baseline on parent stress at 2 months
  Assessment of parent stress
Barkley Deficit in Executive Functions Scale | Change from baseline on parent executive functioning at 2 months
  We will use the Barkley Deficits in Executive Functioning Scale for Adults (BDEFS; Barkley, 2011) which is an empirically based tool for evaluating dimensions of adult executive functioning in daily life. We will use the Overall Executive Functioning Total Score which is a sum of all 89 items (each rated on a likert scale from 1 "never or rarely" to 4 "very often" such that higher scores represent greater degrees of executive functioning impairments) and possible values on the Total Score range from 89 to 356.
Child and Adolescent Symptom Inventory (CASI-V) | Change from baseline on ADHD and oppositional behaviors at 2 months
  Assessment of ADHD and oppositional behaviors
Strengths and Difficulties Questionnaire | Change from baseline on child impairments at 2 months
  Assessment of child impairments

CONTACTS AND LOCATIONS:
Overall Officials: Linda Pfiffner, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- HALP Clinic, Children's Center at Langley Porter, UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No